CLINICAL TRIAL: NCT01310764
Title: Efficacy and Safety of Trabeculectomy With Subconjunctival Bevacizumab Versus Trabeculectomy With Mitomycin C.
Brief Title: Trabeculectomy With Subconjunctival Bevacizumab Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rassoul Akram Hospital (Other)
Responsible Party: Naveed Nilforushan, Rassoul Akram Hospital,Ophthalmic Research Center,Department of Ophthalmology,Iran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 971
Record Dates: First submitted 2011-03-07; First posted 2011-03-08 (Estimated); Last update posted 2011-03-29 (Estimated); Status verified 2009-04

CONDITIONS: Glaucoma
Keywords: Intraocular pressure; Trabeculectomy; Mitomycin C; Bevacizumab
MeSH Terms: conditions — Glaucoma | interventions — Trabeculectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mitomycin C (Sham Comparator): Those with trabeculectomy and intraoperative application of mitomycin C.
  Interventions: Procedure: Trabeculectomy
- Bevacizumab (Active Comparator): Those with trabeculectomy and adjunctive intraoperative subconjunctival injection of bevacizumab.
  Interventions: Procedure: Trabeculectomy

INTERVENTIONS:
Procedure: Trabeculectomy — Both groups underwent trabeculectomy ,but in active group bevacizumab was used and in sham group mitomycin c was used during the surgery.

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of bevacizumab as an adjunctive treatment to trabeculectomy in open angle glaucoma patients and to compare this new drug to the most commonly used anti-scarring agent, mitomycin C.

DETAILED DESCRIPTION:
The most common surgical technique for controlling the intraocular pressure in glaucoma patients is trabeculectomy.In this surgery, internal cavity of the eye is connected by a fistula like openings to subconjunctival space. The main cause of failure in trabeculectomy is excessive postoperative conjunctival scarring at the site of fistula, which is related to severity of conjunctival vascularization, tortuousity of vessel, and fibroblast migration and proliferation. At the time of surgery most surgeons use mitomycin C, which is an antimitotic and antifibrotic agent, to improve the results of the procedure. Although this agent is very effective, but is not without complication. The most significant and sight threatening complications are low intraocular pressure and endophthalmitis. Therefore investigations are going on to find a much safer and effective agents. Bevacizumab is a monoclonal antibody against vascular endothelial factor (VEGF). VEGF is an important vasculogenic and fibrogenic factor with a prominent role in wound healing.Bevacizumab is widely used in ophthalmology and has a promising effect in treatment of neovascularization in conjunctiva, cornea and retina. There are limited animal and human case series regarding the effect of this agent in trabeculectomy. In this study the investigators are trying, in addition to evaluating the efficacy and safety of this agent in result of trabeculectomy, compare this agent with mitomycin C.

ELIGIBILITY:
Inclusion Criteria:

* Uncontrolled Open angle glaucoma.
* Glaucoma patients who are non-compliant to medical treatment.
* Progressive glaucoma despite of medical treatment.
* Follow-up of at least 6 months after surgery

Exclusion Criteria:

* History of prior ocular surgery.
* Pregnancy or breast feeding.
* Age < 18 years.
* History of ocular surface infection in recent two weeks.
* History of systemic thrombo-embolic events.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-04; Primary Completion 2009-11 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure. | 7-12 months
  Pre and post operative intraocular pressures are measured with Goldmann applanation tonometer at each time point visits and the measurement were compared between both groups.

SECONDARY OUTCOMES:
Number of medications. | 7-12 months
  Number of pre and post operative medications were recorded and compared in each post operative visits.

CONTACTS AND LOCATIONS:
Locations (1):
- Rassoul Akram hospital, eye research center, Tehran, Tehran Province, Iran

REFERENCES:
- [Background] Grewal DS, Jain R, Kumar H, Grewal SP. Evaluation of subconjunctival bevacizumab as an adjunct to trabeculectomy a pilot study. Ophthalmology. 2008 Dec;115(12):2141-2145.e2. doi: 10.1016/j.ophtha.2008.06.009. Epub 2008 Aug 9. PMID 18692246
- [Background] Memarzadeh F, Varma R, Lin LT, Parikh JG, Dustin L, Alcaraz A, Eliott D. Postoperative use of bevacizumab as an antifibrotic agent in glaucoma filtration surgery in the rabbit. Invest Ophthalmol Vis Sci. 2009 Jul;50(7):3233-7. doi: 10.1167/iovs.08-2441. Epub 2009 Jan 31. PMID 19182254